CLINICAL TRIAL: NCT04046367
Title: Prehabilitation in Bariatric Surgery: a Randomized Controlled Clinical Trial
Brief Title: Prehabilitation in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Insular Gran Canaria (Other)
Collaborators: Fundación MAPFRE Guanarteme (Unknown)
Responsible Party: Principal Investigator, Rosa María Sánchez Hernández, Attending Physician, Hospital Universitario Insular Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-170
Record Dates: First submitted 2019-06-14; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: nutrition; physical activity; prehabilitation
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Preoperative Exercise; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial, which will compare two group interventions in patients on the waiting list for bariatric surgery.
  Duration: 4-month intervention, with biweekly 2-hour group sessions c / un, followed by a monthly reinforcement session of 1h until surgical intervention.
  Intervention A: Educational program and cognitive-behavioral intervention (group control) Intervention B: Educational program and cognitive-behavioral intervention, with specific training aimed at increasing physical activity, capacity functional and conditioning of the respiratory musculature (group of intervention).
Who Masked: Participant, Outcomes Assessor
Masking Description: A person external to the monitoring and evaluation of the patients will generate a random sequence (by computer), to assign the participants to their corresponding treatment group. The intervention sequence will be transcribed to cards that will be introduced in an envelope each. The envelopes will be opaque, sealed and numbered consecutively. Each time a patient agrees to participate in the trial, he/she signs the informed consent and we verify that he/she meets the inclusion criteria, but not the exclusion criteria, the corresponding envelope will be opened in correlative order.
  Patients will be assigned to one of two group interventions, unaware of the components in each group. The assessment of most of the outcomes will be blinded, too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Educational program and cognitive-behavioral intervention. The patient receives training in nutrition and cognitive-behavioral therapy, with specific training aimed at increasing physical activity, functional capacity and conditioning of the respiratory musculature (prehabilitation by a physiotherapist)
  Interventions: Behavioral: Prehabilitation
- Control (Active Comparator): Educational program and cognitive-behavioral intervention. The patient receives training in nutrition and cognitive-behavioral therapy, as well as standard instructions to increase physical activity.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Prehabilitation — Prehabilitation: The intervention of a physiotherapist will be added to the components of the control group. Patients will receive practical instructions on aerobic and resistance physical activity, as well as training of their inspiratory muscles.
  Other Names: Inspiratory muscle training, physical activity.
  Arms: Intervention
Behavioral: Control — Standard group intervention. Educational program and cognitive-behavioral intervention. The patient receives training in nutrition and cognitive-behavioral therapy, as well as standard instructions to increase physical activity.
  Arms: Control

SUMMARY:
Obesity is a major public health problem in our region and constitutes a priority of the Canary Islands Health Plan. Bariatric surgery is the most effective intervention in the treatment of obesity and its complications. However, people with obesity have high surgical risk and long-term outcomes are related to pre-surgical weight loss.

In patients currently on the bariatric surgery waiting list, a randomized controlled trial will be performed in which two group interventions will be compared. One of the interventions (standard), will consist of educational modules in food and exercise, combined with cognitive-behavioral therapy. In the other, a specific training (prehabilitation) will be added to encourage physical activity and the conditioning of inspiratory muscles.

The pre-surgical weight loss (principal outcome) will be compared between groups, as well as the evolution of the complications of obesity, the functional status of the patients, their physical activity, quality of life, immediate complications of surgery and days of admission.

DETAILED DESCRIPTION:
Obesity is a major public health problem, responsible for an increased risk of hypertension, obesity, dyslipidemia, type 2 diabetes, cardiovascular disease, some types of cancer, psychiatric diseases and mortality.

Bariatric surgery has proven to be the most effective method for reducing weight and related comorbidities in patients with morbid obesity. However, pre-surgical weight loss reduces postsurgical complications. In addition, weight loss before surgery seems to be the only factor positively associated with post-surgical weight loss, and this effect seems to be more pronounced in patients with BMI> 45 kg / m2.

Pre-operative physical conditioning (prehabilitation) can improve the patient's functional capacity before major surgery. Most studies showing this have been conducted in orthopedic surgery and abdominal cancer surgery. There are very few studies that evaluate prehabilitation in patients undergoing bariatric surgery.

Objective

Comparison of a multidisciplinary group intervention with another one to which specific training focused on increasing physical activity is added, in patients on the surgical waiting list for bariatric surgery in a randomized controlled trial.

Methods

Design Randomized, controlled parallel group, clinical trial.

Intervention Duration: 4-month intervention, with biweekly 2,5-hour group sessions, followed by a monthly reinforcement session of 1h until surgery.

Intervention A: Educational program and cognitive-behavioral intervention (control group)

Intervention B: Educational program and cognitive-behavioral intervention, with specific training aimed at increasing physical activity, functional capacity and conditioning of the respiratory muscles (intervention group).

Study population The recruitment of the participants will be made from the waiting list of bariatric surgery (obesity II-IV), selecting patients with estimated waiting time above 4 months. Patients will be excluded if any reason for inadequate follow-up is identified, according to the investigators criteria.

Ethical aspects The design and execution of this study will be done in accordance with the Declaration of Helsinki and the homogenized European guidelines of good clinical practice. Before their participation, the patients will sign an informed consent form. The protocol has been approved by the local ethics committee

Sample size Based on the size of the waiting list for bariatric surgery, with a mean duration of 17 months, and that the intervention is considered feasible on two groups of 10 people, in parallel, in each branch, (a weekly session of 2h per nutrition nurse, with support from additional professional). Starting with a pilot group of each intervention and taking into account an overlap between them, in 18 months about 60-80 patients could be included in total.

With 80 patients included, without losses, and assuming a standard deviation of weight of 11Kg, and for a bilateral p <0.05 a difference between groups of 7 and 8Kg, with a statistical power of 80 and 90%, respectively. If we assume a standard deviation of 6Kg, as shown by other studies, the detectable difference would be reduced to about 4Kg.

Statistical analysis A descriptive analysis of the baseline situation will be made. The qualitative variables are expressed as a percentage, quantitative, as mean (SD) or median, according to if its distribution is normal or not, respectively. Comparisons will be made between treatment groups, using chi squared for qualitative variables and Student's t or Mann Whitney's U for quantitative variables. The analysis of results will be done by intention to treat analysis. That is, all patients who have baseline data and have been randomized, will be included, regardless of their subsequent attendance to the Program.

ELIGIBILITY:
Inclusion Criteria:

* People with obesity (type II-IV), on the waiting list for bariatric surgery in the Complejo Hospitalario Universitario Materno-infantil de Las Palmas

Exclusion Criteria:

* any factor that, in the opinion of the researchers, limits the ability to monitor the intervention (language barrier, ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-22 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | 4-6 months
  Increase (or decrease) in weight between the start of the program and the time of surgery (measured on a calibrated scale, with Maximum increments of 0.1Kg, under the same conditions, without footwear and with light clothing)

SECONDARY OUTCOMES:
Body mass index | 4-6 months
  Calculated as weight (in Kg) divided by the squared height (in meters)
Body composition | 4-6 months
  Percentage of body fat and lean mass estimated by bioimpedance
Associated complications-Blood pressure | 4-6 months
  Systolic and diastolic blood pressure (in sitting position, after 5 minutes of rest, using a manual sphygmomanometer, with a cuff adapted to thebrachial circumference of the patient)
Associated complications-lipids | 4-6 months
  total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides (automatic methods) in mg/dl colorimetric tests)
Associated complications-glucose metabolism | 4-6 months
  HbA1c (HPLC standardized against DCCT-IFCC)
Associated complications-treatments | 4-6 months
  Number of drugs used for associated cardiovascular risk factors
Associated complications-liver enzymes | 4-6 months
  AST, ALT, GGT (automatic methods)
Adherence to the intervention | 4-6 months
  Attendance at the sessions (number of sessions attended) programmed.
Physical activity-steps | 4-6 months
  Registered by pedometers (number of steps/week)
Physical activity-self reported | 4-6 months
  International Physical Activity Program (IPAQ) questionnaire
Eating patterns-Adherence to Mediterranean diet | 4-6 months
  Validated Food questionnaire (simplified questionnaire of 14 questions of adherence to the diet Mediterranean diet of PREDIMED) . Higher scores indicate higher adherence
Eating patterns-eating disorders | 4-6 months
  Standardised questionnaire (bulimia and binge disorders of the EDI -Eating Disorder Inventory)
General health status | 4-6 months
  EQ-5D questionnaire (higher scores indicate better self-perceived health status)
Emotional state | 4-6 months
  Hospital scale of anxiety and depression (HADS)
Subjective evaluation of satisfaction, perceived effort and motivation | 4-6 months
  Development of a specific questionnaire with Likert type scale for the patient to score 1 to 10 each of the 3 items.
Functional capacity-walk test | 4-6 months
  6-minute walk test (TM6): meters completed during the test
Functional capacity- grip strength | 4-6 months
  Grip test: hand grip dynamometer and the grip strength in both hands, indicating the dominant one.
Functional capacity-respiratory muscle strength | 4-6 months
  Maximum inspiratory pressure (PIM) and expiratory pressure (PEM)
Functional capacity-plethysmography | 4-6 months
  Lung volumes, VR (residual volume) and CRF (functional residual capacity) in ml
Functional capacity-Spirometry | 4-6 months
  Forced spirometry: Forced expiratory volume in 1 second (FEV1), Functional Vital Capacity (FVC) in ml. Tiffenau index will be calculated. Mesoespiratory flows
Functional capacity-sleep apnea questionnaire | 4-6 months
  Stop-bang screening questionnaire for sleep-related breathing disorders.
Functional capacity-sleep apnea polygraph | 4-6 months
  Home cardiorespiratory polygraphy for diagnosis of disorder
Surgical complications | 5-7 months after start of intervention
  Early post-surgical complications (<30 days)
Surgery-length of admission | 5-7 months after start of intervention
  Post-surgical length of stay (stratified by surgical technique).

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Wägner, MD, PhD, Principal Investigator — Complejo Hospitalario Universitario Insular Materno-Infantil de Gran Canaria
Locations (1):
- Complejo Hospitalario Universitario Materno-infantil de Las Palmas, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the results
Access Criteria: Reasonable plan, acknowledgement of original investigators